CLINICAL TRIAL: NCT03793010
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of FX006 in Patients With Hip Osteoarthritis
Brief Title: Study to Evaluate the Efficacy and Safety of FX006 in Patients With Hip Osteoarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: By Sponsor due to occurrences of incomplete study drug administration
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2018-015
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Results first posted 2020-09-14 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Hip
Keywords: Osteoarthritis; Hip; Pain; Intra-articular; Injection
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Pain | interventions — FX006; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FX006 (Experimental): FX006 32mg
  Interventions: Drug: FX006
- Normal Saline (Placebo Comparator): Normal Saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: FX006 — Single Intra-articular injection
  Arms: FX006
Drug: Normal saline — Single Intra-articular injection
  Arms: Normal Saline

SUMMARY:
This is a two-part, multi-center, randomized, double-blind, placebo-controlled, parallel-group study in patients with hip OA. Approximately 70 patients will be enrolled in Part I and approximately 440 patients will be enrolled in Part II of the study. In each part, patients will be randomized to one of two treatment groups (1:1) and treated with a single IA injection of either 32 mg FX006 or normal saline.

DETAILED DESCRIPTION:
This is a two-part, multi-center, randomized, double-blind, placebo-controlled, parallel-group study in patients with hip OA. Approximately 70 patients will be enrolled in Part I and approximately 440 patients will be enrolled in Part II of the study. In each part, patients will be randomized to one of two treatment groups (1:1) and treated with a single IA injection of either 32 mg FX006 or normal saline.

FX006 or saline placebo will be administered as a single IA injection with a 12-week follow-up period in the double-blind phase.

Patients participating in Part I of the study will be treated with a single IA injection of either 32 mg FX006 or normal saline and will return for follow up visits at Weeks 12, 16, 20, and 24. The patients will be discontinued at the time of notification by the Investigator.

Patients participating in Part II of the study will be treated with a single IA injection of either 32 mg FX006 or normal saline and will return for follow up visits at Weeks 12, 16, 20, and 24.

Patients participating in Part II of the study that are not clinically indicated for a second injection at Week 12 will return to the clinic at Weeks 16, 20, and 24 and will receive an open-label injection of FX006 at the first evaluation where the patient has been determined to meet all criteria. Patients will then return for follow-up visits every 4 weeks for 12 weeks post second injection and will complete the study 12 weeks post second injection (e.g., Week 24, 28, 32, or 36 depending on when the patient receives the open-label injection).

Patients participating in Part II of the study who are not eligible for a second injection after evaluation at Weeks 12, 16, 20, and 24 will complete the study at the Week 24 visit and complete the End of Study (EOS) assessments.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Patients 40 to 80 years of age, inclusive, on the day of randomization (Day 1)
* Body Mass Index (BMI) ≤ 40 kg/m2
* Symptoms associated with OA of the index hip for ≥ 3 months prior to Screening visit
* Currently meet the American College of Radiology (ACR) Criteria (clinical and radiological) for OA of the index hip
* Kellgren-Lawrence (KL) Grade 2 or 3 in the index hip as confirmed by X-ray during Screening visit (centrally read)
* Qualifying mean score on the WOMAC A and C (0-10 NRS scale)
* Agree to maintain the similar activity level throughout the study
* Willingness to abstain from use of restricted medications

Exclusion Criteria:

* Patients who cannot washout of prohibited medications
* Diagnosed as secondary OA in the index hip including but not limited to articular fracture, major dysplasia or congenital abnormality, osteochondritis dissecans, acromegaly, ochronosis, hemochromatosis, Wilson's disease, or primary osteochondromatosis, etc.
* Ipsilateral chronic knee pain
* Sciatica
* Atrophic osteoarthritis, femoral head necrosis and/or collapse, or subchondral bone insufficiency fracture in the index hip joint determined via central reading
* Current or history of infection in the index hip (e.g. osteomyelitis) or current skin infection at injection site
* Trauma or surgeries (e.g., arthroscopy, knee surgery) of lower limbs within 52 weeks with sequelae, etc.
* History or current evidence of reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease, systemic lupus erythematosus or other autoimmune diseases
* Any planned surgeries in the lower limbs during the study period, or any other surgery during the study period that would require use of a restricted medication
* Presence of surgical hardware or other foreign body in the index hip
* Planned/anticipated surgery of the index hip or any other surgery that would require use of a restricted medication during the study period
* IA corticosteroid of any joint within 3 months of Screening visit (investigational or marketed, including FX006)
* IA treatment of index hip with any of the following agents within 6 months of Screening: any biologic agent or hyaluronic acid (investigational or marketed)
* IV or IM corticosteroids (investigational or marketed) within 3 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening visit
* Planned or expected changes to lifestyle with regard to physical activity, physical therapy, acupuncture, transcutaneous electrical nerve stimulation (TENS), or bracing within 1 month prior to Screening and changes throughout the duration of the study
* Women of child-bearing potential (not surgically sterile or post-menopausal for at least 1 year as documented in medical history) not using a highly effective method or who are pregnant or nursing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (32):
- United States (32):
  - Arizona Research Center, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - TriWest Research Associates, LLC, El Cajon, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Tampa Bay Medical Research, Clearwater, Florida
  - Florida Research Associates, LLC, DeLand, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Medallion Clinical Research Institute, LLC, Naples, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - National Pain Research Institute, Winter Park, Florida
  - Better Health Clinical Research, Inc, Newnan, Georgia
  - Injury Care Research, LLC, Boise, Idaho
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Heartland Research Associates, Newton, Kansas
  - Excel Clinical Research, Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Charleston, South Carolina
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Spectrum Medical, Inc., Danville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was from December 2018 until August 2019. The patients were enrolled at medical clinics.
Period: Overall Study
Arm/Group | FX006 | Normal Saline
Started | 35 | 35
Randomized But Not Dosed | 2 | 0
Completed | 7 | 8
Not Completed | 28 | 27
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Withdrawn by Investigator or Sponsor | 19 | 18
Not completed — Lost to Follow-up | 1 | 2
Not completed — Patient couldn't sit still for injection | 1 | 0
Not completed — Withdrew to pursue other treatment | 1 | 0
Not completed — Did not meet eligibility criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received a full dose of study drug assigned to the FX006 32 mg arm and the placebo arm were included in the analysis. 68 total patients were included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | FX006 | Normal Saline | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.45) | 61.8 (7.99) | 60.7 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 28 | 31 | 59
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 24 | 26 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 33 | 35 | 68
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.50 (5.679) | 31.29 (5.775) | 30.91 (5.699)

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC A (Pain) Score at Week 12
Description: The change from baseline on the average Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A (pain) score at Week 12. The average WOMAC A score is calculated by taking the average of five questions with a range from 0 (no pain) to 10 (extreme pain).
Time Frame: Baseline and Week 12
Population: All patients who received a full dose of study drug assigned to the FX006 32 mg arm and the placebo arm were included in the analysis. 68 total patients were included in the safety analysis. 55 of 68 patients had Week 12 assessments and are included in the primary and secondary outcomes analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FX006 | Normal Saline
Number analyzed (Participants) | 24 | 31
score on a scale | -1.85 [-2.99 to -0.71] | -2.16 [-3.22 to -1.09]
Statistical Analysis 1: Comparison: FX006 vs Normal Saline; Test type: Superiority; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-1.20 to 1.81]

2. Secondary Outcome: Change in WOMAC C (Function) Score at Week 12
Description: Change from Baseline on the WOMAC C (function) score at Week 12. The average WOMAC C score is calculated by taking the average of seventeen questions with a range from 0 (no difficulty) to 10 (extreme difficulty).
Time Frame: Baseline and Week 12
Population: All patients who received a full dose of study drug assigned to the FX006 32 mg arm and the placebo arm were included in the analysis. 68 total patients were included in the safety population. 55 of 68 patients had week 12 assessments and are included in the primary and secondary outcomes analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FX006 | Normal Saline
Number analyzed (Participants) | 24 | 31
score on a scale | -1.56 [-2.73 to -0.40] | -2.16 [-3.30 to -1.03]
Statistical Analysis 1: Comparison: FX006 vs Normal Saline; Test type: Superiority; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-1.05 to 2.24]

3. Secondary Outcome: PGIC Score at Week 12
Description: PGIC (Patient Global Impression of Change) at Week 12. The PGIC score has a range from 1(very much improved) to 7 (very much worse) and indicates the overall status of the patient since baseline.
Time Frame: 12 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FX006 | Normal Saline
Number analyzed (Participants) | 24 | 31
score on a scale | 3.4 [2.7 to 4.1] | 3.4 [2.8 to 4.1]
Statistical Analysis 1: Comparison: FX006 vs Normal Saline; Test type: Superiority; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-1.0 to 0.9]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for FX006 32 mg and Placebo from Baseline to Last Visit at Week 24.
Arm/Group | FX006 | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 21/33 | 14/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FX006 (N=33) | Normal Saline (N=35)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 1
Adhesion (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Repetitive Strain Injury (Injury, poisoning and procedural complications) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Blood Pressure Diastolic Increased (Investigations) | 1 | 1
Blood Pressure Increased (Investigations) | 2 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0
Weight Increased (Investigations) | 2 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Decreased Apetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 2 | 0
Renal Cyst (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor due to occurrences of incomplete study drug administration. Only 15% of the planned study population had enrolled and no statistical evaluations reported due to insufficient sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT03793010/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03793010/SAP_001.pdf